CLINICAL TRIAL: NCT01156818
Title: Wheezometer™ Exploratory (WM) Field Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KarmelSonix Ltd. (Industry)
Responsible Party: Ross Wilson, KarmelSonix
Other Study IDs: KSI-MUL-GEN-WMF-01
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2010-07

CONDITIONS: Respiratory Sounds; Wheezing
Keywords: Wheeze measurements
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children: Age 8-21 years
- Adult: Age 21-80 years

SUMMARY:
Karmel Sonix Ltd has developed the Personal WheezoMeter a hand-held pulmonary sounds analyzer that utilizes contact sensors to acquire, amplify, filter, record and quantify the presence of wheezing. When used to monitor conditions such as asthma, this device should be used under the direction of a physician or licensed healthcare professional. The device is intended for use with pediatric and adult patients in both home and clinical settings.

The purpose of the study is to determine whether Wz% and change in Wz% correlate with symptoms and change in symptoms at least as well as FEV1 and change in FEV1.0. Additional information to be obtained from the study will be to determine whether there is a symptom threshold at which a patient seeks rescue medications and if so, to determine the value of Wz% and FEV1.0 at this point (Wz%, FEV1.0 thresholds). The study will also provide information on the within patient and whole group correlations between Wz% and FEV.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed asthma.
* Poorly controlled asthma as per GINA Guidelines with frequent (i.e. >5/week) use of reliever medications.
* Adequate comprehension level and demonstrated ability to perform unsupervised spirometry, wheezometry and use the symptom diary.
* Age range 8-80. Patients over 40 will only be included if they are lifetime non-smokers, who have demonstrated reversibility of airway obstruction (at least 12% improvement in FEV1.0 after bronchodilator).
* All patients included in the study will be routinely receiving either a short acting bronchodilator or a long acting bronchodilator twice daily as part of their regular medication. Additional doses of bronchodilator will be taken on an as needed basis. No change in regular medication will be made for the purposes of the study.
* Subject or subject's parents/guardians is/are able to comprehend and give informed consent for participation in the study.

Consent of treating physician.

Exclusion Criteria:

* Inability to perform spirometry and/or Wheezometry. Skin Disorder (burn, infection, or allergy) over upper chest (Child) or neck (Adult).
* Patients with other diseases, which in the opinion of the treating physician would interfere with the management of asthma and performance of the study according to the protocol.
* Hospitalization at recruitment, [patients who get admitted while participating will continue to participate].

P- hysician objection.

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Asthma patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Wz% change in response to BD. Symptom score by e-Diary; Spirometer - FEV1.0/FVC/PEF/MEF50 with automated storage and timing | 2 weeks

SECONDARY OUTCOMES:
Correlate Wz% to FEV1.0: within patient correlation | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ross Wilson, Study Director — KarmlSonix
Locations (1):
- California Allergy and Asthma Medical Group, Inc., Los Angeles, California, United States